CLINICAL TRIAL: NCT07273500
Title: Precision Exercise Prescription for Obese Children With Bronchial Asthma: a Dose-dependent Study on Adiposity Biomarkers, Body Composition, and Respiratory Efficiency
Brief Title: Precision Exercise in Obese Children With Bronchial Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0023/041
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-10

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: A prospective, three-arm, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: A single-blind protocol was adopted. The researcher who collected the data was blind to the allocation of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): The control group completed the 12-week respiratory re-training program alongside a moderate-intensity aerobic regimen (50-70% of maximum heart rate), maintaining a total weekly exercise volume not exceeding 75 minutes.
  Interventions: Other: Respiratory Re-training
- Low-dose group (Experimental): For the low-dose condition, participants engaged in the standard respiratory re training and supplemental aerobic exercise at 50-70% of maximum heart rate, capping the cumulative weekly duration at 150 minutes across the 12-week intervention.
  Interventions: Other: Low-dose Aerobic Training
- High-dose group (Experimental): The high-dose group performed the core respiratory re-training in addition to a moderate-intensity aerobic regimen (50-70% of maximum heart rate), which was systematically escalated to a maintenance volume of 300 minutes per week throughout the 12-week trial.
  Interventions: Other: High-dose Aerobic Training

INTERVENTIONS:
Other: Respiratory Re-training — The standardized respiratory re-training protocol was administered in 30-minute sessions, three times per week, over a consecutive 12-week period. The regimen incorporated diaphragmatic breathing, breath-holding and control techniques, pursed-lip breathing, respiratory muscle strengthening, postural correction, and relaxation exercises.
  Arms: Control group
Other: Low-dose Aerobic Training — A moderate-intensity aerobic regimen (50-70% of maximum heart rate) maintained at a consistent total weekly volume of 150 minutes.
  Arms: Low-dose group
Other: High-dose Aerobic Training — A moderate-intensity aerobic regimen (50-70% of maximum heart rate) maintained at a consistent total weekly volume of 300 minutes.
  Arms: High-dose group

SUMMARY:
This investigation recruited 72 pediatric patients with a confirmed bronchial asthma diagnosis. Participants were randomized into three cohorts: a control group undertaking under 75 minutes of weekly aerobic activity, a low-dose group completing 150 minutes/week, and a high-dose group performing 300 minutes/week. Exercise intensity was maintained between 50-70% of the age- adjusted maximum heart rate across 3-4 supervised sessions per week for a 12-week intervention period.

Pre- and post-intervention analyses included measurements of adipose-tissue- derived adipokines, circulating inflammatory markers, body composition, and pulmonary function parameters.

DETAILED DESCRIPTION:
Study Population and Recruitment

A total of 72 pediatric patients with bronchial asthma were enrolled from the Pulmonary Medicine/Critical Care and Allergy-Immunology departments of King Khalid Hospital and two additional tertiary care centers in Riyadh, Saudi Arabia. Eligible participants were children aged 8 to 18 years with a diagnosis of moderate, clinically stable BA and a body mass index ranging from 30.0 to 35.0 kg/m². Further inclusion criteria stipulated the absence of lower limb or spinal deformities, stable medication regimens for the preceding three months, and no participation in structured physical activity for at least six months prior to the study. Exclusion criteria encompassed acute exacerbation of asthma symptoms, the presence of other chronic pulmonary diseases, and any pre- existing cardiovascular or musculoskeletal disorder that could impede exercise training.

Outcome Measures

Adiposity and Inflammatory Biomarkers: Serum concentrations of key adipokines-specifically total adiponectin, high-molecular-weight adiponectin, leptin, and resistin-were analyzed. Concurrently, systemic inflammatory mediators, including interleukin-6 and high-sensitivity C-reactive protein, were quantified using commercially available enzyme-linked immunosorbent assay kits.

Body Composition Analysis: A multi-frequency bioelectrical impedance analysis (BIA) device was employed to determine body composition indices. The parameters assessed included body fat percentage, fat mass, fat-free mass, total body water, and basal metabolic rate.

Pulmonary Function Testing: Spirometric evaluations were conducted with a calibrated spirometer to measure forced expiratory volume in one second (FEV1) and forced vital capacity (FVC). The FEV1/FVC ratio was subsequently calculated from these values.

Intervention Protocol

All participants underwent a standardized respiratory re-training program for 12 consecutive weeks. This intervention was administered in 30-minute sessions, three times per week, and comprised diaphragmatic breathing, breath-holding and control exercises, pursed-lip breathing, inspiratory muscle strengthening, postural correction, and relaxation techniques.

Participants were then allocated into three distinct groups, each receiving an additional, varying dose of aerobic training superimposed on the core respiratory program:

Control Group: This group performed supplemental aerobic exercise at a moderate intensity (50-70% of age-predicted maximum heart rate) for a consistent total of less than 75 minutes per week, spread across three sessions.

Low-Dose Group: This cohort engaged in aerobic training at the same moderate intensity, with a target cumulative duration of 150 minutes per week. The duration was progressively increased from a baseline of 90 minutes in the first week by 30 minutes each subsequent week, stabilizing at the target dose by the third week.

High-Dose Group: This group followed the same moderate-intensity aerobic protocol but with a target weekly volume of 300 minutes. A similar progressive ramp-up was implemented, starting at 90 minutes weekly and increasing by 30 minutes per week until the target was achieved in the eighth week, after which it was maintained.

ELIGIBILITY:
Inclusion Criteria:

* Age of 8-18 years
* Body mass index ranging from 30 to 35 kg/m2
* Verified asthma diagnosis per the Global Initiative for Asthma (GINA) criteria
* Moderate Onset
* Clinically Stable
* Maintained medication dosages in the past three months
* Free of lower limb or spinal deformities
* Not engaging in regular exercise regimens in the past six months.

Exclusion Criteria:

* Exacerbated asthma symptoms
* Chronic lung comorbidities
* Cardiovascular or musculoskeletal conditions expected to hinder the training.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2023-09-17 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Leptin | 2 months
  Serum leptin concentration was evaluated as a primary adipokine. It was assayed using a commercially available enzyme-linked immunosorbent assay kit, with pre- and post-training results expressed in nanograms per milliliter (ng/mL).
Total Adiponectin | 2 months
  Serum total adiponectin concentration was quantified as a key adiposity biomarker, pre- and post-training. It was measured using a commercially available enzyme-linked immunosorbent assay kit, with results reported in micrograms per milliliter (µg/mL)
High-molecular-weight Adiponectin | 2 months
  The serum concentration of the high-molecular-weight isoform of adiponectin was analyzed pre- and post-training. It was quantified using a commercial enzyme-linked immunosorbent assay, with levels reported in micrograms per milliliter (µg/mL).
Resistin | 2 months
  Serum resistin concentration was assessed as an adipokine of interest. Levels were determined from pre- and post-training blood samples using a commercial enzyme-linked immunosorbent assay kit, with concentrations reported in nanograms per milliliter (ng/mL).
Interleukin-6 | 2 months
  Systemic concentration of the inflammatory cytokine interleukin 6 was evaluated. Pre- and post-training levels were quantified using a commercially available enzyme-linked immunosorbent assay kit, with results reported in picograms per milliliter (pg/mL).
High-sensitivity C-reactive protein | 2 months
  Systemic concentration of high-sensitivity C-reactive protein was assessed as a marker of low-grade inflammation. Pre- and post-training levels were quantified using a commercially available enzyme-linked immunosorbent assay kit, with results reported in milligrams per liter (mg/L).
Body fat percentage | 2 months
  Body fat percentage was evaluated as a key body composition metric. Pre- and post-training measurements were conducted using a bioelectrical impedance analysis device, with results expressed as a percentage (%).
Fat Mass | 2 months
  Total body fat mass was assessed as a component of body composition. It was measured pre- and post-intervention using a bioelectrical impedance analysis device, with values reported in kilograms (kg).
Fat-free mass | 2 months
  Fat-free mass was evaluated as an indicator of lean body tissue. Pre- and post-training measurements were obtained using a bioelectrical impedance analysis device, with results recorded in kilograms (kg).
Total body water | 2 months
  Total body water was quantified as a fundamental body composition parameter. Pre- and post-training measurements were conducted using a bioelectrical impedance analysis device, with results expressed in liters (L).
Basal Metabolic Rate | 2 months
  Basal metabolic rate was estimated as a measure of resting energy expenditure. Pre- and post-training assessments were conducted using a bioelectrical impedance analysis device, with results reported in kilocalories per day (kcal/day).
Forced Expiratory Volume in One Second | 2 months
  Forced expiratory volume in one second (FEV#) was assessed as a primary spirometric parameter of airway function. Pre- and post-training measurements were obtained using a calibrated spirometer, with results expressed as a percentage of the predicted value (% pred) based on established reference standards.
Forced Vital Capacity | 2 months
  Forced vital capacity (FVC) was evaluated as a key measure of lung volume. Pre- and post-training assessments were performed using a calibrated spirometer, with results expressed as a percentage of the predicted value (% pred).
Forced Expiratory Volume in One Second (FEV1) / Forced Vital Capacity (FVC) Ratio | 2 months
  The ratio of forced expiratory volume in one second to forced vital capacity (FEV1/FVC) was calculated as an indicator of airflow limitation. This derived value was determined from pre- and post-training spirometric maneuvers and is expressed as a ratio (decimal value).

CONTACTS AND LOCATIONS:
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No